CLINICAL TRIAL: NCT05616858
Title: Safety and Cardiopulmonary Efficacy of Complex Exercise Program for Stroke Patients in the Community
Brief Title: Complex Exercise Program for Stroke Patients
Acronym: CEPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sung-Hwa Ko, Associate professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PNUYH_ETRI_2
Record Dates: First submitted 2022-10-31; First posted 2022-11-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Sports Physical Therapy; Program, Communication
MeSH Terms: conditions — Stroke; Communication

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group with exercise program
  Interventions: Behavioral: Complex exercise program
- Control group (No Intervention): Group without exercise program

INTERVENTIONS:
Behavioral: Complex exercise program — Stretching exercise, aerobic exercise, strengthening and balancing exercise
  Arms: Intervention group

SUMMARY:
The physical and social effects of exercise programs and daily exercise have already been demonstrated in stroke. However, stroke survivors have shown a passive attitude towards the exercise program and there was little guideline and experience of the stroke exercise program in the community. Therefore, the study provides patients with an adequate guide to a complex exercise program after discharge based on the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Community indwelling stroke patients discharged from Pusan National University Yangsan Hospital
* Independent ambulator (FAC over 4)
* Independent daily activities (Modified Rankin Scale less than 2)
* No apparent spasticity on hemiplegic side (Modified Ashworth scale less than 1)
* Hemiplegic side motor grades (Manual muscle testing, MMT) more than 3

Exclusion Criteria:

* MMSE less than 18
* BBS less than 41
* Severe aphagia who cannot communicate
* Severe cardiovascular conditions inhibiting exercise programs
* Musculoskeletal problems inhibiting exercise programs
* Other medical conditions considered by physiatrists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | Baseline evaluation
  Maximal VO2 from cardiopulmonary exercise test
Peak VO2 | Follow-up evaluation (through study completion, an average of 6 weeks)
  Maximal VO2 from cardiopulmonary exercise test

SECONDARY OUTCOMES:
Functional ambulation category (0-5, the higher the better) | Baseline evaluation
  6-point functional walking test that evaluates ambulation ability
Functional ambulation category (0-5, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  6-point functional walking test that evaluates ambulation ability
Berg balance scale (0-56, the higher the better) | Baseline evaluation
  Objectively determine a patient's ability to safely balance during a series of predetermined tasks
Berg balance scale (0-56, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Objectively determine a patient's ability to safely balance during a series of predetermined tasks
Timed up and go | Baseline evaluation
  To determine fall risk and measure the progress of balance
Timed up and go | Follow-up evaluation (through study completion, an average of 6 weeks)
  To determine fall risk and measure the progress of balance
Grip strength | Baseline evaluation
  measure of muscular strength or the maximum force/tension generated by one's forearm muscles
Grip strength | Follow-up evaluation (through study completion, an average of 6 weeks)
  measure of muscular strength or the maximum force/tension generated by one's forearm muscles
6-minute walk test | Baseline evaluation
  practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians
6-minute walk test | Follow-up evaluation (through study completion, an average of 6 weeks)
  practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians
Figure-of-eight walk test | Baseline evaluation
  Measurement tool that assesses the ability to walk on a curved path
Figure-of-eight walk test | Follow-up evaluation (through study completion, an average of 6 weeks)
  Measurement tool that assesses the ability to walk on a curved path
Sit-and-reach test | Baseline evaluation
  Measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles
Sit-and-reach test | Follow-up evaluation (through study completion, an average of 6 weeks)
  Measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles
Chair sit-to-stand test | Baseline evaluation
  Testing leg strength and endurance in older adults
Chair sit-to-stand test | Follow-up evaluation (through study completion, an average of 6 weeks)
  Testing leg strength and endurance in older adults
Fugl-Meyer assessment (0-226, the higher the better) | Baseline evaluation
  Stroke-specific, performance-based impairment index
Fugl-Meyer assessment (0-226, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Stroke-specific, performance-based impairment index
Manual function test (0-32, the higher the better) | Baseline evaluation
  Evaluate unilateral manual performance in hemiparetic patients after stroke
Manual function test (0-32, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Evaluate unilateral manual performance in hemiparetic patients after stroke
Modified Barthel Index (Korean version) (0-100, the higher the better) | Baseline evaluation
  Measure of physical disability used widely to assess behaviour relating to activities of daily living
Modified Barthel Index (Korean version) (0-100, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Measure of physical disability used widely to assess behaviour relating to activities of daily living
Body composition analysis | Baseline evaluation
  Percentage of fat, bone, and muscle in the body
Body composition analysis | Follow-up evaluation (through study completion, an average of 6 weeks)
  Percentage of fat, bone, and muscle in the body
Korean Mini-Mental Status Examination (K-MMSE) (0-30, the higher the better) | Baseline evaluation
  Screening of dementia and to investigate the possible changes of optimal cutoff scores
Korean Mini-Mental Status Examination (K-MMSE) (0-30, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Screening of dementia and to investigate the possible changes of optimal cutoff scores
Euro-Quality of Life-5 Dimension (EQ-5D) (5-25, the higher the better) | Baseline evaluation
  A brief and simple instrument measuring health related quality of life
Euro-Quality of Life-5 Dimension (EQ-5D) (5-25, the higher the better) | Follow-up evaluation (through study completion, an average of 6 weeks)
  A brief and simple instrument measuring health related quality of life
Getriatic depression scale (0-15, the higher the more depressive) | Baseline evaluation
  Assessment of depression in the elderly
Getriatic depression scale (0-15, the higher the more depressive) | Follow-up evaluation (through study completion, an average of 6 weeks)
  Assessment of depression in the elderly
International Physical Activity Questionnaire (No scores) | Baseline evaluation
  27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old
International Physical Activity Questionnaire (No scores) | Follow-up evaluation (through study completion, an average of 6 weeks)
  27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No